CLINICAL TRIAL: NCT02776059
Title: A Phase II, Multicenter, Randomized, Open-label Study to Investigate the Safety and Efficacy of Pegfilgrastim (Neulasta®) in Patients With Alcoholic Hepatitis
Brief Title: Pegfilgrastim in Patients With Alcoholic Hepatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Timothy Morgan, MD (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor-Investigator, Timothy Morgan, MD, Chief of Hepatology, Southern California Institute for Research and Education
Organization: Southern California Institute for Research and Education (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCAH Consortium- AH Treatment; 5U01AA021886 (NIH)
Record Dates: First submitted 2016-05-10; First posted 2016-05-18 (Estimated); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Alcoholic Hepatitis
Keywords: survival; pegfilgrastim; cirrhosis, alcoholic
MeSH Terms: conditions — Hepatitis, Alcoholic; Liver Cirrhosis, Alcoholic | interventions — Standard of Care; pegfilgrastim; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- prednisolone or pentoxifylline + pegfiltrastim (Experimental): prednisolone or pentoxifylline for 28 days PO plus pegfilgrastim subcutaneous weekly shot
  Interventions: Drug: Standard of care + pegfiltrastim
- prednisolone or pentoxifylline (Active Comparator): prednisolone or pentoxifylline for 28 days
  Interventions: Drug: Standard of care

INTERVENTIONS:
Drug: Standard of care + pegfiltrastim — prednisolone or pentoxifyline orally for 28 days + pegfilgrastim (Neulasta®) 6 mg in 0.6 mL SQ
  Other Names: Neulasta®
  Arms: prednisolone or pentoxifylline + pegfiltrastim
Drug: Standard of care — Oral prednisolone or pentoxifyline for 28 days only
  Other Names: prednisolone or pentoxifyline
  Arms: prednisolone or pentoxifylline

SUMMARY:
This is a multi-center, prospective, randomized trial of standard of care vs. standard of care + pegfilgrastim (Neulasta®) among patients with a clinical diagnosis of alcoholic hepatitis and DF≥32.

DETAILED DESCRIPTION:
Standard of care treatment will be with either prednisolone 40 mg/day for 28 days or pentoxifylline 400 mg TID for 28 days. The patient's physician will decide the standard of care treatment the patient will receive. Patients will be randomized (1:1) to receive either no additional drug treatment (SOC group) or to receive a pegfilgrastim (Neulasta®, 6 mg) SQ.

Patients will be seen in-person at screening, randomization (Day 1), Day 8, Day 29, Week 12, and Week 24. Safety examination and blood tests will be performed. In addition, biological specimens will be saved for research purposes at these time points.

Total duration of patient participation is 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of alcoholic hepatitis with Maddrey's discriminant function score ≥32. Age 18 years or older.

Exclusion Criteria:

* Renal failure (creatinine >2.0 mg/dl)
* Bilirubin <5 mg/dL
* uncontrolled recent upper gastrointestinal bleeding
* Known HIV infection
* Uncontrolled infection, or pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-01-21 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Adverse events, especially infection and renal failure, Change in MELD Score and DF between Day 1 and Day 29, Lille score (at Day 8) | Day 1, Day 8, Day 29, and Day 90
  The primary outcome will be survival at Day 90. Assuming a fixed sample size of 70 patients (35 per arm), a one-sided z-test will have 81.6% power to detect a 25% improvement in survival proportions between arms, with survival in the standard of care arm at 65%.

SECONDARY OUTCOMES:
adverse events | 24 weeks
  adverse events through Week 24
Liver function | Day 29
  Change in MELD and Maddrey DF during first 4 weeks
liver function | Day 8
  Change in Lille score
Survival | at Day 90
  survival at Day 90

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Morgan, MD, Study Chair — VA Long Beach Healthcare System
Locations (5):
- United States (5):
  - VA Loma Linda Healthcare System, Loma Linda, California
  - VA Long Beach Healthcare System, Long Beach, California
  - LAC-USC Medical Center, Los Angeles, California
  - Harbor-UCLA Medical Center, Torrance, California
  - New Mexico VA Health Care System, Albuquerque, New Mexico

IPD SHARING:
Plan to Share IPD: Yes
Patients' coded data will be shared .

REFERENCES:
- [Derived] Tayek JA, Stolz AA, Nguyen DV, Fleischman MW, Donovan JA, Alcorn JM, Chao DC, Asghar A, Morgan TR; Southern California Alcoholic Hepatitis (SCAH) Consortium. A phase II, multicenter, open-label, randomized trial of pegfilgrastim for patients with alcohol-associated hepatitis. EClinicalMedicine. 2022 Oct 12;54:101689. doi: 10.1016/j.eclinm.2022.101689. eCollection 2022 Dec. PMID 36267499